CLINICAL TRIAL: NCT03458273
Title: Multi-center, Observational, Retrospective Comparison of the Feasibility, Safety, and Efficacy of Real Zero Fluoroscopy Versus Conventional Fluoroscopic Catheter Ablation With and Without 3D System Support: Propensity Matched Study
Brief Title: Real Zero Fluoroscopy Catheter Ablation.
Acronym: ZERO-Fluoro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Maciej Wójcik, MD, PhD, Associate Professor, Medical University of Lublin
Other Study IDs: MW-MULublin-2
Record Dates: First submitted 2018-02-24; First posted 2018-03-08 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Atrial Arrhythmia; Ventricular Arrythmia; Arrhythmia; Arrhythmias, Cardiac
Keywords: Atrial Arrhythmia; Ventricular Arrythmia; ablation; fluoroscopy
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Zero fluoro: Patients in whom Zero fluoroscopy ablation was performed under the guidance of Ensite for mapping and ablation and fluoroscopy will not be used during the procedure.
  Interventions: Procedure: Zero fluoroscopy ablation
- Conventional ablation without 3D: Patients in whom Conventional fluoroscopy ablation was performed under fluoroscopic guidance only.
  Additional use of Ensite/Carto/Localisa for mapping was not allowed.
  Interventions: Procedure: Conventional ablation without 3D
- Conventional ablation with 3D: Patients in whom Conventional fluoroscopy ablation was performed under fluoroscopic and Ensite/Carto guidance and ablation during the procedure.
  Use of fluoroscopy and additional Ensite/Carto for mapping and ablation was mandatory.
  Interventions: Procedure: Conventional ablation with 3D

INTERVENTIONS:
Procedure: Zero fluoroscopy ablation — Catheter ablation for the treatment of atrial and ventricular arrhythmia - no fluoroscopy guidance
  Other Names: Zero fluoro
  Groups: Zero fluoro
Procedure: Conventional ablation without 3D — Catheter ablation for the treatment of atrial and ventricular arrhythmia - fluoroscopy guidance only. 3D system (Every Ensite/Carto) is not allowed
  Other Names: Conventional fluoroscopy ablation without 3D
  Groups: Conventional ablation without 3D
Procedure: Conventional ablation with 3D — Catheter ablation for the treatment of atrial and ventricular arrhythmia - fluoroscopy guidance + 3D system support (Ensite/Carto)
  Other Names: Conventional fluoroscopy ablation with 3D
  Groups: Conventional ablation with 3D

SUMMARY:
A Retrospective Propensity Matched Study comparing:

* real zero fluoroscopy catheter ablation
* conventional fluoroscopy catheter ablation without 3D system
* conventional fluoroscopy catheter ablation with 3D system

DETAILED DESCRIPTION:
Catheter ablation is a well-established treatment to treat patients with a wide scope of heart arrhythmias.

The study is an investigator-initiated, retrospective analysis of prospectively collected data. The study population consists of patients with right-sided arrhythmias who underwent zero-fluoroscopy catheter ablation between the years 2016 and 2018 in 3 centers and a propensity score matched patients group of patients who:

* underwent conventional fluoroscopy guided catheter ablation without 3D system (Ensite/Carto) support
* underwent conventional fluoroscopy guided catheter ablation with 3D system (Ensite/Carto) support

Covariates for matching will be:

* arrhythmia type
* age of a patient
* number of diagnostic catheters used during a procedure
* type of a diagnostic catheter used during a procedure]

ELIGIBILITY:
Inclusion Criteria:

* right atrial tachycardia
* right atrial premature complexes
* AVNRT
* right atrial AVRT/WPW
* right ventricle tachycardia / right ventricle premature complexes

Exclusion Criteria:

* left atrium arrhythmia
* left ventricle arrhythmia

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Zero fluoroscopy group: patients after right atrium/ventricle arrhythmia ablation performed with 3D (Ensite/Carto) guidance but without fluoroscopy guidance
  Convectional fluoroscopy group: patients after right atrium/ventricle arrhythmia ablation performed with fluoroscopy guidance but without 3D (Ensite/Carto) guidance
  Convectional fluoroscopy group + 3D: patients after right atrium/ventricle arrhythmia ablation performed with fluoroscopy guidance and with 3D (Ensite/Carto) guidance
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Procedural success rates | 3 months
  arrhythmia recurrence within 3 months since the index procedure

SECONDARY OUTCOMES:
Total procedure time | during procedure
  total procedure time measured as needle to needle time
Fluoroscopy time | during procedure
  total fluoroscopy time during procedure
Acute procedural success | 10-30 minutes
  acute procedural success defined as arhhythia elimination
Recurrence rate | 6 months
  arrhythmia recurrence within 6 months since the index procedure
Acute Complications rate | during procedure
  Procedural Complications procedure
All Complications rate | 6 months
  Procedural Complications and Complications within 6 months since the index procedure
The length of stay during the hospitalization | 1 month
  Number of hospital days for ablation procedure from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Wójcik, MD, PhD, Principal Investigator — Medical University of Lublin, Poland
Locations (3):
- Poland (3):
  - Wojewódzki Szpital Specjalistyczn, Biała Podlaska
  - Medical University of Lublin, Lublin
  - SP ZOZ Szpital Puławy, Puławy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang L, Sun G, Chen X, Chen G, Yang S, Guo P, Wang Y, Wang DW. Meta-Analysis of Zero or Near-Zero Fluoroscopy Use During Ablation of Cardiac Arrhythmias. Am J Cardiol. 2016 Nov 15;118(10):1511-1518. doi: 10.1016/j.amjcard.2016.08.014. Epub 2016 Aug 24. PMID 27639689
- [Background] Casella M, Ribatti V, Catto V, Vettor G, Fassini G, Biagioli V, Dello Russo A, Tondo C. Benefits of electroanatomic ablation of conventional cardiac arrhytmias: from fluoroscopy to zero X-ray mapping. Minerva Cardioangiol. 2018 Feb;66(1):49-62. doi: 10.23736/S0026-4725.17.04478-4. Epub 2017 Aug 31. PMID 28862408
- [Background] Gaita F, Guerra PG, Battaglia A, Anselmino M. The dream of near-zero X-rays ablation comes true. Eur Heart J. 2016 Sep 21;37(36):2749-2755. doi: 10.1093/eurheartj/ehw223. Epub 2016 Jun 26. PMID 27354053
- [Background] Seizer P, Bucher V, Frische C, Heinzmann D, Gramlich M, Muller I, Henning A, Hofbeck M, Kerst G, Gawaz M, Schreieck J. Efficacy and safety of zero-fluoroscopy ablation for supraventricular tachycardias. Use of optional contact force measurement for zero-fluoroscopy ablation in a clinical routine setting. Herz. 2016 May;41(3):241-5. doi: 10.1007/s00059-015-4358-4. Epub 2015 Oct 13. PMID 26462477
- [Background] Bulava A, Hanis J, Eisenberger M. Catheter Ablation of Atrial Fibrillation Using Zero-Fluoroscopy Technique: A Randomized Trial. Pacing Clin Electrophysiol. 2015 Jul;38(7):797-806. doi: 10.1111/pace.12634. Epub 2015 Apr 16. PMID 25790320
- [Background] Scaglione M, Ebrille E, Clemente FD, Gaita F, Bradfield JS. Catheter Ablation of Atrial Fibrillation Without Radiation Exposure Using A 3D Mapping System. J Atr Fibrillation. 2015 Feb 28;7(5):1167. doi: 10.4022/jafib.1167. eCollection 2015 Feb-Mar. PMID 27957146
- [Result] Alvarez M, Bertomeu-Gonzalez V, Arcocha MF, Morina P, Tercedor L, Ferrero de Loma A, Pachon M, Garcia A, Pardo M, Datino T, Alonso C, Osca J; investigators of the Spanish Multicenter Registry of Fluoroscopy-free Ablation. Nonfluoroscopic Catheter Ablation. Results From a Prospective Multicenter Registry. Rev Esp Cardiol (Engl Ed). 2017 Sep;70(9):699-705. doi: 10.1016/j.rec.2016.12.040. Epub 2017 Jan 31. English, Spanish. PMID 28159569